CLINICAL TRIAL: NCT04880096
Title: Constitution and Analysis of a Cohort of Patients Followed in Pain Clinics and at Home in Real Life
Brief Title: Cohort of Chronic Pain Patients
Acronym: e-DOL cohort
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut ANALGESIA (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 AUTHIER
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; e-Health
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic pain patients: All adult patients followed-up in participating pain clinics
  Interventions: Other: eDOL

INTERVENTIONS:
Other: eDOL — e-health tool (mobile app for patients and web platform for caregivers in pain clinics)

SUMMARY:
Chronic pain affects approximately 20% of adults, 50% of the elderly population and over 1.5 billion people worldwide. Societal and economic issues are also crucial, as 60% of people with pain are less able or unable to work and 20% say they have lost their jobs because of pain. The overall cost of chronic pain is estimated at around 300 billion euros in the EU. Unfortunately, current treatments for chronic pain have limited effectiveness and important adverse effects. Pain clinics, which support the most complex and refractory cases of chronic pain, as well as general practitioners and patients expect improvements, both in terms of therapeutic efficacy and organization of care.

In order to allow the characterization and a personalized follow-up of chronic pain patients, we have created e-DOL, a smartphone application for patients and a web platform for healthcare professionals in pain clinics. The purpose of this study is to create an e-cohort for the research, and characterization and follow-up of chronic pain patients.

DETAILED DESCRIPTION:
This first French e-cohort of chronic pain patients will allow real-life follow-up in order to generate big data including various information on chronic pain, associated-comorbidities, pain impacts on sleep, activity and psycho-emotional parameters, sociodemographic characteristics and pain treatments.

These data will be collected with he eDOL tool (smartphone application for patients and web platform for caregivers in pain clinics), integrating numerous repeatable questionnaires, weekly barometers, a therapeutic education module and a conversational agent (chat bot).

All of these data will also be linked with French health insurance care data in order to get an overview of comorbidities and patient care consumption in a medico-economic approach.

The study will include 20 pain clinics and a minimum of 5000 patients followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients with chronic pain
* patients equipped and regular users of a smartphone
* Non-opposition to participation in the study

Exclusion Criteria:

* Patient unable to understand or answer questionnaires

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patiant with chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
multidimensional characterisation of chronic pain patients | 5 years
  Multimodal exploratory analysis of the determinants and repercussions of chronic pain, and their evolution in a real-life context, taking into account all environmental events likely to influence chronic pain (treatments, history, co-morbidities, etc.).

SECONDARY OUTCOMES:
Multivariate descriptive analyses | 5 years
  Study the relationships between the measured criteria
Longitudinal analyses | 5 years
  Describe the distribution and temporal evolution of the measured variables

CONTACTS AND LOCATIONS:
Locations (22):
- France (22):
  - CHU de Clermont-Ferrand - Service de Neurologie, Clermont-Ferrand, AURA
  - Clermont-Ferrand University Hospital, Clermont-Ferrand, AURA
  - APHP Ambroise Paré, Boulogne-Billancourt, IDF
  - APHP Saint Antoine, Paris, IDF
  - APHP Cochin, Paris, IDF
  - Groupe Hospitalier Paris Saint Joseph, Paris, IDf
  - CHU Amiens, Amiens
  - CH Bayeux, Bayeux
  - CHU bordeaux, Bordeaux
  - Hospices civils Lyon, Bron
  - CHU Grenoble, Grenoble
  - CHU Limoges, Limoges
  - Ch Lons Le Saunier, Lons-le-Saunier
  - CHU Montepllier, Montpellier
  - CHU Nantes, Nantes
  - CHU Nîmes, Nîmes
  - CHU Rennes, Rennes
  - Chu Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Hôpital Civil de Strasbourg, Strasbourg
  - Chu Toulouse, Toulouse
  - CH Voiron, Voiron

REFERENCES:
- [Derived] Delage N, Cantagrel N, Soriot-Thomas S, Frost M, Deleens R, Ginies P, Eschalier A, Corteval A, Laveyssiere A, Phalip J, Bertin C, Pereira B, Chenaf C, Doreau B, Authier N; ePAIN; Kerckhove N. Mobile Health App and Web Platform (eDOL) for Medical Follow-Up of Patients With Chronic Pain: Cohort Study Involving the French eDOL National Cohort After 1 Year. JMIR Mhealth Uhealth. 2024 Jun 12;12:e54579. doi: 10.2196/54579. PMID 38865173